CLINICAL TRIAL: NCT02772939
Title: Evaluation of Arterial Stiffness as a Predictor of Response to Renal Sympathetic Denervation
Brief Title: Arterial Stiffness as a Predictor of Response to Renal Sympathetic Denervation
Acronym: EFFECTIVENES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Effectiveness0001
Record Dates: First submitted 2016-03-10; First posted 2016-05-16 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Therapy Resistant Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation (Experimental): Renal denervation for therapy resistant arterial hypertension
  Interventions: Device: Renal sympathetic denervation (RDN)

INTERVENTIONS:
Device: Renal sympathetic denervation (RDN) — Catheter based renal sympathetic denervation for therapy resistant arterial hypertension

SUMMARY:
This trial is designed to establish invasive and non-invasive measures of arterial stiffness as potential predictors of treatment response to renal sympathetic denervation

DETAILED DESCRIPTION:
Regardless of the ongoing debate on the general effect of renal sympathetic denervation in therapy resistant hypertension, all trials published so far face the problem of a certain proportion of nonresponders to treatment. Previous data shows, that to some extent this might be attributable to arterial stiffening. Elevated invasive pulse wave velocity as an established marker for arterial stiffness has been found to be associated with nonresponse to renal denervation treatment in a smaller trial population. This trial attempts to assess the predictive value of different invasive and non-invasive markers for arterial stiffness in an adequately powered population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with therapy resistant arterial hypertension (>=3 antihypertensive drugs including at least one diuretic without any dosage change in the preceding 4 weeks) and office BP >160 mmHg systolic or 90 mmHg diastolic

Exclusion Criteria:

* average systolic daytime BP <135 mmHg in 24h ambulatory blood pressure measurement (ABPM)
* pregnancy
* known renal artery stenosis
* >= 1 renal artery diameter < 4 mm
* life expectancy <6 months
* participation in any other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2020-09 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Predictive value of invasive Pulse wave velocity for blood pressure response after renal denervation | 3 Months
  difference in daytime blood pressure (ABPM) between patients with low (<14.4 m/s) vs. high invasive pulse wave velocity
Predictive value of noninvasive and invasive measures of arterial stiffness (Pulse wave velocity assessed invasively, with a piezoelectric device and MRI-based) in combination with clinical variables | 3 Months
  AUC of ROCs for noninvasive and invasive measures of arterial stiffness in predicting blood pressure response to renal denervation

SECONDARY OUTCOMES:
Change in 24h ambulatory blood pressure | 3 months, 6 months, 12 months
Change in exercise blood pressure | 3 months
Predictive value of MRI-assessed aortic distensibility on Change in daytime ambulatory blood pressure | 3 months, 6 months, 12 months
Predictive value of MRI-assessed aortic distensibility on Change in 24 h ambulatory blood pressure | 3 months, 6 months, 12 months
Predictive value of MRI-assessed total arterial compliance on Change in daytime ambulatory blood pressure | 3 months, 6 months, 12 months
Predictive value of MRI-assessed total arterial compliance on Change in 24 h ambulatory blood pressure | 3 months, 6 months, 12 months
comparison of predictive value of invasive pulse wave velocity, invasive central pulse pressure, noninvasive pulse wave velocity, noninvasive central pulse pressure, aortic distensibility, total arterial compliance for Change in ambulatory blood pressure | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No